CLINICAL TRIAL: NCT06684665
Title: Introduction;Epidemiology;Socioeconomic Burden
Brief Title: Study on the Sociopsychoemotional Mechanism of Dysfunction in Patients With Acute and Chronic Low Back Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-13-219
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy group: The healthy subjects were subjects without back pain
- Acute low back pain group: The acute low back pain group was defined as those with low back pain that lasted less than three months
- Chronic low back pain group: The chronic low back pain group was the subjects with low back pain, and the duration was greater than or equal to three months

SUMMARY:
Low back pain is defined as pain that extends from the 12th rib to the iliac bone, and its increasing incidence makes it one of the major causes of decreased productivity worldwide. Dysfunction is one of the important complications in patients with chronic low back pain, and related studies have shown that depression, pain catastrophization and other emotions can affect the occurrence and development of dysfunction. So the investigators wanted to study which psychological emotions affect the development of dysfunction in patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75;
2. Patients with low back pain;
3. Have good communication skills to ensure the collection of scale information

Exclusion Criteria:

1. Suffering from severe mental or psychiatric disorders.;
2. Unwilling to participate in the interview;
3. Patients with pain in other areas

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients who met the requirements of outpatient complaints and healthy people in daily life
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Dysfunction index of patients with acute and chronic low back pain | From enrollment to 2 months later
  Dysfunction is one of the important complications in patients with chronic low back pain, and related studies have shown that depression, pain catastrophization and other emotions can affect the occurrence and development of dysfunction. The dysfunction index of patients with different course of disease was different from that of healthy people.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China